CLINICAL TRIAL: NCT07141810
Title: Early Antifibrotic Therapy for f-ILD
Brief Title: Efficacy and Safety of Early Antifibrotic Therapy for Non-progressive Fibrotic Interstitial Lung Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jiuwu Bai, Doctor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025022295
Record Dates: First submitted 2025-02-28; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Fibrotic Interstitial Lung Disease
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: One group was treated with basic therapy alone, and another group was treated with basic therapy combined with antifibrotic therapy.
Who Masked: Investigator
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antifibrotic drug (Active Comparator)
  Interventions: Drug: Antifibrotic drugs (nidanib or pirfenidone)
- Primary therapy group (No Intervention): One group received primary therapy，without antifibrotic drug

INTERVENTIONS:
Drug: Antifibrotic drugs (nidanib or pirfenidone) — One group received primary therapy, and another group received an antifibrotic drug (nidanib or pirfenidone) in addition to primary therapy.
  Arms: Antifibrotic drug

SUMMARY:
Early antifibrotic therapy for f-ILD

ELIGIBILITY:
Inclusion Criteria:

1) Able to understand the procedures and methods of this study, willing to strictly follow the clinical trial protocol to complete this study, and sign the informed consent; 2) The age of signing the informed consent is 40-85 years old (including both ends of the value); 3) Weight: male ≥50 kg, female ≥40 kg; 4) During screening, FVC accounted for more than 45% of the estimated value and 90%; 5) The percentage of pulmonary carbon monoxide dispersion (DLCO) to the predicted value (corrected by Hb value) during screening was ≥30% and ≤90%; 6) Diagnosed with fibrotic ILD: In the past 12 months, at least 3 months after basic treatment such as glucocorticoids and immunosuppressants, reexamination of chest CT showed fibrotic features such as diffuse mesh shadow, honeycomb lung, and tractive bronchiectasis in both lungs, and the lesions could not be further absorbed.

-

Exclusion Criteria:

1. Patients with unstable disease (IPF) assessed by investigators during screening had acute exacerbations during screening or within 3 months before randomization;
2. Patients who are likely to require lung transplantation within 6 months or whose expected survival is less than 1 year as assessed by the investigators at the time of screening;
3. During screening, chest HRCT indicated that the range of emphysema exceeded the range of pulmonary fibrosis (based on independent imaging evaluation results);
4. Patients with airway obstruction disease (such as FEV1/FVC after bronchodilator);
5. Diagnosed with IPF
6. Diagnosis of PPF according to the 2022 ATS/ERS/JRS/ALAT guidelines
7. Patients with other types of respiratory diseases that the investigators assessed might affect the study results;
8. Patients who need to receive oxygen therapy for 15 hours or more per day;
9. Resting pulse oxygen < 90% (sea level to 1500m above sea level) or < 85% (altitude > 1500m) when breathing indoor air during screening;
10. with other poorly controlled underlying conditions (such as NYHA Class III or IV congestive heart failure, acute myocardial infarction, unstable angina, hemorrhagic or ischemic stroke, pulmonary hypertension requiring treatment within the 6 months prior to screening), Patients assessed by the investigator as unsuitable for the study;
11. Patients who had an active tuberculosis infection in the 12 months prior to screening, or had a bacterial, viral, fungal, or microbial infection requiring treatment with any clinical symptoms within the 4 weeks prior to randomization;
12. Patients diagnosed with NCOV infection 1 month before screening and/or during screening (NCOV nucleic acid testing is not part of this study and can be performed on demand);
13. Patients who plan to receive NCOV vaccine and other vaccines from 1 month before screening to 1 month after the last dose;
14. Patients with a history of malignant tumors (except cured basal cell carcinoma of the skin and cervical carcinoma in situ) within 5 years prior to screening, or who are currently being evaluated for potential malignant tumors;
15. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 upper limit of normal (ULN) or total bilirubin ≥1.5× upper limit of normal (ULN);
16. Serum creatinine ≥1.5× upper limit of normal (ULN);
17. Active hepatitis, syphilis or HIV antibody positive patients;
18. Major surgery (general anesthesia) within 3 months prior to screening, or surgery planned to be performed during the study period that the investigator assessed would affect the study endpoint;
19. Participated in any clinical trial (including other investigational drug/investigational device therapy) within 3 months prior to screening, or was still within 5 half-lives of the investigational drug at the time of screening;
20. Current smoking history, smoking cessation ≤3 months, or unable to abstain from smoking for the entire study period;
21. Suspected or confirmed history of alcohol or drug abuse;
22. Known allergy to the investigational drug and its ingredients;
23. Pregnant and lactating women, female subjects who plan to become pregnant during the study period, or patients who do not wish to use contraceptives that meet the protocol requirements during the trial;
24. Other conditions assessed by the investigator as unsuitable for participation in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
FVC %predict | 48 weeks

IPD SHARING:
Plan to Share IPD: Undecided